CLINICAL TRIAL: NCT03189719
Title: A Randomized, Double-Blind, Placebo-Controlled Phase III Clinical Trial of Pembrolizumab (MK-3475) in Combination With Cisplatin and 5-Fluorouracil Versus Placebo in Combination With Cisplatin and 5-Fluorouracil as First-Line Treatment in Subjects With Advanced/Metastatic Esophageal Carcinoma (KEYNOTE-590)
Brief Title: First-line Esophageal Carcinoma Study With Pembrolizumab Plus Chemo vs. Chemo (MK-3475-590/KEYNOTE-590)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3475-590; 173739 (Registry Identifier: JAPIC-CTI); MK-3475-590 (Other: MSD); KEYNOTE-590 (Other: MSD); 2017-000958-19 (EudraCT Number)
Record Dates: First submitted 2017-06-14; First posted 2017-06-16 (Actual); Results first posted 2021-07-06 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Esophageal Neoplasms
Keywords: Programmed Cell Death-1 (PD1, PD-1),; Programmed Cell Death Receptor Ligand 1 (PDL1, PD-L1); Programmed Cell Death Receptor Ligand 2 (PDL2, PD-L2)
MeSH Terms: conditions — Esophageal Neoplasms; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab; Cisplatin; Fluorouracil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pembrolizumab + SOC (Experimental): Participants receive pembrolizumab 200 mg intravenously (IV) every 3 weeks (Q3W) plus standard of care (SOC) chemotherapy with cisplatin 80 mg/m^2 IV Q3W and 5-FU 800 mg/m^2/day continuous IV infusion on Days 1 to 5 (120 hours) Q3W. All treatments will be administered on an outpatient basis beginning on Day 1 of each 3-week dosing cycle.
  Interventions: Biological: Pembrolizumab; Drug: Cisplatin; Drug: 5-FU
- Placebo + SOC (Placebo Comparator): Participants receive placebo to pembrolizumab (saline) IV Q3W plus SOC chemotherapy with cisplatin 80 mg/m^2 IV Q3W and 5-FU 800 mg/m^2/day continuous IV infusion on Days 1 to 5 (120 hours) Q3W. All treatments will be administered on an outpatient basis beginning on Day 1 of each 3-week dosing cycle.
  Interventions: Drug: Placebo; Drug: Cisplatin; Drug: 5-FU

INTERVENTIONS:
Biological: Pembrolizumab — 200 mg administered IV Q3W on Day 1 of each 3-week cycle, up to 35 administrations.
  Other Names: MK-3475
  Arms: Pembrolizumab + SOC
Drug: Placebo — Placebo to pembrolizumab (saline) administered IV Q3W on Day 1 of each 3-week cycle, up to 35 administrations.
  Arms: Placebo + SOC
Drug: Cisplatin — 80 mg/m^2 administered IV Q3W on Day 1 of each 3-week cycle. Duration of cisplatin treatment will be capped at 6 doses.
Drug: 5-FU — 800 mg/m^2/day (4000 mg/m^2 total per cycle) administered as continuous IV infusion on Days 1 to 5 (120 hours) of each 3-week cycle, or per local standard for 5-FU administration, up to 35 administrations.

SUMMARY:
The purpose of this trial is to evaluate efficacy and safety of pembrolizumab plus standard of care (SOC) chemotherapy with cisplatin and 5-fluorouracil (5-FU) versus placebo plus SOC chemotherapy with cisplatin and 5-FU as first-line treatment in participants with locally advanced or metastatic esophageal carcinoma.

The overall primary efficacy hypotheses are as follows:

1. In participants with esophageal squamous cell carcinoma (ESCC), participants whose tumors are programmed cell death-ligand 1 (PD-L1)-positive (defined as combined positive score [CPS] ≥10), ESCC participants whose tumors are PD-L1 positive (CPS ≥10), and in all participants, overall survival (OS) is superior with pembrolizumab plus SOC chemotherapy compared with placebo plus SOC chemotherapy.
2. In participants with ESCC, participants whose tumors are PD-L1 positive (CPS ≥10), and in all participants, progression-free survival (PFS) according to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 as assessed by investigator is superior with pembrolizumab plus SOC chemotherapy compared with placebo plus SOC chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Has histologically- or cytologically-confirmed diagnosis of locally advanced unresectable or metastatic adenocarcinoma or squamous cell carcinoma of the esophagus or advanced/metastatic Siewert type 1 adenocarcinoma of the esophagogastric junction (EGJ)
* Has measurable disease per RECIST 1.1 as determined by the local site investigator/radiology assessment
* Eastern Cooperative Group (ECOG) performance status of 0 to 1
* Can provide either a newly obtained or archival tissue sample for PD-L1 by immunohistochemistry analysis
* Female participants of childbearing potential must have a negative urine or serum pregnancy test within 72 hours prior to randomization and be willing to use an adequate method of contraception (e.g. abstinence, intrauterine device, diaphragm with spermicide, etc.) for the course of the study through 120 days after the last dose of study treatment and up to 180 days after last dose of cisplatin
* Male participants of childbearing potential must agree to use an adequate method of contraception (e.g. abstinence, vasectomy, male condom, etc.) starting with the first dose of study treatment through 120 days after the last dose of study treatment and up to 180 days after last dose of cisplatin, and refrain from donating sperm during this period
* Has adequate organ function

Exclusion Criteria:

* Has locally advanced esophageal carcinoma that is resectable or potentially curable with radiation therapy (as determined by local investigator)
* Has had previous therapy for advanced/metastatic adenocarcinoma or squamous cell cancer of the esophagus or advanced/metastatic Siewert type 1 adenocarcinoma of the EGJ
* Has had major surgery, open biopsy, or significant traumatic injury within 28 days prior to randomization, or anticipation of the need for major surgery during the course of study treatment
* Has a known additional malignancy that is progressing or requires active treatment. Exceptions include early-stage cancers (carcinoma in situ or Stage 1) treated with curative intent, basal cell carcinoma of the skin, squamous cell carcinoma of the skin, in situ cervical cancer, in situ breast cancer that has undergone potentially curative therapy, and in situ or intramucosal pharyngeal cancer
* Has known active central nervous system metastases and/or carcinomatous meningitis.
* Has an active autoimmune disease that has required systemic treatment in past 2 years
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study treatment, or has a history of organ transplant, including allogeneic stem cell transplant
* Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis, or has an active infection requiring systemic therapy
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of study medication and up to 180 days after last dose of cisplatin
* Has received prior therapy with an anti-programmed cell death protein-1 (anti-PD-1), anti-PD-L1, or anti-PD-L2 agent or with an agent directed to another co-inhibitory T-cell receptor or has previously participated in a pembrolizumab (MK-3475) clinical trial
* Has severe hypersensitivity (≥ Grade 3) to any study treatment (pembrolizumab, cisplatin, or 5-FU) and/or any of its excipients
* Has a known history of active tuberculosis (TB; Mycobacterium tuberculosis) or human immunodeficiency virus (HIV) infection
* Has known history of or is positive for hepatitis B or hepatitis C
* Has received a live vaccine within 30 days prior to the first dose of study treatment
* Has had radiotherapy within 14 days of randomization. Participants who received radiotherapy >14 days prior to randomization must have completely recovered from any radiotherapy-related AEs/toxicities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 749 (Actual)
Dates: Start 2017-07-25 (Actual); Primary Completion 2020-07-02 (Actual); Study Completion 2023-07-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (189):
- United States (12):
  - Kaiser Permanente Southern California ( Site 0003), West Los Angeles, California
  - The University of Chicago Medical Center ( Site 0001), Chicago, Illinois
  - University of Kansas ( Site 0029), Westwood, Kansas
  - University of Maryland Medical Center ( Site 0013), Baltimore, Maryland
  - Dana Farber Cancer Center ( Site 0009), Boston, Massachusetts
  - Henry Ford Cancer Center ( Site 0018), Detroit, Michigan
  - Washington University School of Medicine ( Site 0031), St Louis, Missouri
  - Roswell Park Cancer Institute ( Site 0004), Buffalo, New York
  - Weill Cornell Medical College ( Site 0024), New York, New York
  - University Hospitals Cleveland Medical Center ( Site 0002), Cleveland, Ohio
  - UPMC Cancer Center/Hillman Cancer Center ( Site 0015), Pittsburgh, Pennsylvania
  - University of Tennessee Medical Center Knoxville ( Site 0017), Knoxville, Tennessee
- Argentina (5):
  - Centro de Investigaciones Clinicas - Clinica Viedma ( Site 0603), Viedma, Río Negro Province
  - Hospital Aleman ( Site 0605), Buenos Aires
  - Hospital Municipal de Gastroenterologia Dr. Bonorino Udaondo ( Site 0602), Buenos Aires
  - Sanatorio Allende - Cordoba ( Site 0604), Córdoba
  - Hospital Privado Centro Medico Cordoba ( Site 0601), Córdoba
- Australia (5):
  - Blacktown Hospital ( Site 2000), Blacktown, New South Wales
  - Liverpool Hospital. ( Site 2001), Liverpool, New South Wales
  - Princess Alexandra Hospital ( Site 2005), Woolloongabba, Queensland
  - Eastern Health ( Site 2002), Box Hill, Victoria
  - Peter MacCallum Cancer Centre ( Site 2003), Melbourne, Victoria
- Brazil (10):
  - CETUS Hospital Dia Oncologia ( Site 0208), Belo Horizonte, Minas Gerais
  - Inst de Medicina Integral Professor Fernando Figueira- IMIP ( Site 0210), Recife, Pernambuco
  - Instituto Nacional do Cancer Jose Alencar Gomes da Silva INCA ( Site 0209), Rio de Janeiro, Rio de Janeiro
  - Hospital Sao Vicente de Paulo ( Site 0204), Passo Fundo, Rio Grande do Sul
  - Uniao Brasileira de Educacao e Assistencia Hospital Sao Lucas da Pucrs ( Site 0201), Porto Alegre, Rio Grande do Sul
  - Clinica de Hematologia e Oncologia Viver Ltda ( Site 0211), Santa Maria, Rio Grande do Sul
  - Fundacao Faculdade Regional de Medicina de Sao Jose do Rio Preto. ( Site 0203), São José do Rio Preto, São Paulo
  - Hospital Alemao Oswaldo Cruz ( Site 0207), São Paulo, São Paulo
  - Hospital de Clinicas de Porto Alegre ( Site 0200), Porto Alegre
  - Instituto do Cancer de Sao Paulo - ICESP ( Site 0206), São Paulo
- Canada (8):
  - Tom Baker Cancer Centre ( Site 0503), Calgary, Alberta
  - Cross Cancer Institute ( Site 0502), Edmonton, Alberta
  - CancerCare Manitoba ( Site 0500), Winnipeg, Manitoba
  - Juravinski Cancer Center ( Site 0508), Hamilton, Ontario
  - The Ottawa Hospital - Cancer Care ( Site 0501), Ottawa, Ontario
  - Princess Margaret Cancer Centre ( Site 0505), Toronto, Ontario
  - CISSS de la Monteregie-Centre ( Site 0504), Greenfield Park, Quebec
  - Jewish General Hospital ( Site 0507), Montreal, Quebec
- Chile (4):
  - Hospital Regional de Concepcion Dr. Guillermo Grant Benavente ( Site 1003), Concepción
  - Pontificia Universidad Catolica de Chile ( Site 1001), Santiago
  - Hospital Clinico Universidad de Chile ( Site 1002), Santiago
  - Clinica Alemana de Temuco ( Site 1006), Temuco
- China (19):
  - Anhui Provincial Hospital ( Site 0106), Hefei, Anhui
  - The First Affiliated Hospital of Anhui Medical University ( Site 0112), Hefei, Anhui
  - Peking Union Medical College Hospital ( Site 0123), Beijing, Beijing Municipality
  - The First Affiliated Hospital of Xiamen University ( Site 0119), Xiamen, Fujian
  - Guangdong General Hospital ( Site 0103), Guangzhou, Guangdong
  - The Affiliated Tumour Hospital of Harbin Medical University ( Site 0102), Harbin, Heilongjiang
  - Tongji Medical College Huazhong University of Science and Technology ( Site 0109), Wuhan, Hubei
  - Hunan Cancer Hospital ( Site 0105), Changsha, Hunan
  - PLA Cancer Centre of Nanjing Bayi Hospital ( Site 0110), Nanjing, Jiangsu
  - Zhongda Hospital Southeast University ( Site 0125), Nanjing, Jiangsu
  - Jilin Cancer Hospital ( Site 0101), Changchun, Jilin
  - The First Affiliated Hospital of Xi an Jiaotong University ( Site 0120), Xi'an, Shannxi
  - Zhejiang Cancer Hospital ( Site 0116), Hangzhou, Zhejiang
  - Beijing Cancer Hospital ( Site 0100), Beijing
  - Fujian Provincial Cancer Hospital ( Site 0104), Fuzhou
  - Shanghai Chest Hospital ( Site 0111), Shanghai
  - Fudan University Shanghai Cancer Center ( Site 0108), Shanghai
  - Renji Hospital Shanghai Jiaotong University School of Medicine ( Site 0114), Shanghai
  - Henan Cancer Hospital ( Site 0107), Zhengzhou
- Colombia (2):
  - Rodrigo Botero SAS ( Site 2703), Medellín, Antioquia
  - Oncomedica S.A. ( Site 2701), Montería, Departamento de Córdoba
- Costa Rica (3):
  - CIMCA Centro de Investigacion y Manejo del Cancer ( Site 2600), San José
  - Policlinico San Bosco ( Site 2602), San José
  - ICIMED - Instituto de Investigacion en Ciencias Medicas ( Site 2601), San José
- Denmark (2):
  - Rigshospitalet ( Site 2301), Copenhagen
  - Odense Universitetshospital ( Site 2300), Odense
- France (8):
  - Centre Leon Berard ( Site 0307), Lyon, Cedex 8
  - CHU Brest - Institut de Cancerologie et d Hematologie ( Site 0305), Brest
  - Centre Francois Baclesse ( Site 0310), Caen
  - Centre Oscar Lambret ( Site 0304), Lille
  - Institut du Cancer de Montpellier ( Site 0306), Montpellier
  - CHU de Nantes - Hotel Dieu ( Site 0303), Nantes
  - Institut Mutualiste Montsouris ( Site 0300), Paris
  - CHU de Saint Etienne Hopital Nord ( Site 0309), Saint-Etienne
- Germany (7):
  - Staedtisches Klinikum Dresden ( Site 1507), Dresden
  - Haematologisch-Onkologische Praxis Eppendorf Facharztzentrum Eppendorf - Hope ( Site 1502), Hamburg
  - Universitaetsklinikum Leipzig ( Site 1501), Leipzig
  - Klinikum Ludwigsburg ( Site 1509), Ludwigsburg
  - Universitatsklinikum Mannheim GmbH ( Site 1504), Mannheim
  - Klinik fuer Haematologie. Onkologie und Gastroenterologie ( Site 1508), Mönchengladbach
  - III. Medizinische Klinik Klinikum rechts der Isar ( Site 1506), München
- Guatemala (5):
  - Centro de Investigacion Oncologica ( Site 1402), Guatemala City
  - Oncomedica ( Site 1400), Guatemala City
  - Grupo Medico Angeles ( Site 1401), Guatemala City
  - Medi-K Cayala ( Site 1404), Guatemala City
  - Centro Regional de Sub Especialidades Medicas SA ( Site 1403), Quetzaltenango
- Hong Kong (4):
  - Humanity Health Research Centre ( Site 1603), Hong Kong
  - Pamela Youde Nethersole Eastern Hospital ( Site 1601), Hong Kong
  - Princess Margaret Hospital. ( Site 1602), Hong Kong
  - Queen Mary Hospital ( Site 1600), Hong Kong
- Japan (31):
  - Aichi Cancer Center Hospital ( Site 0902), Nagoya, Aichi-ken
  - National Cancer Center Hospital East ( Site 0908), Kashiwa, Chiba
  - National Hospital Organization Shikoku Cancer Center ( Site 0901), Matsuyama, Ehime
  - Hokkaido University Hospital ( Site 0916), Sapporo, Hokkaido
  - Hyogo Cancer Center ( Site 0913), Akashi, Hyōgo
  - Kobe City Medical Center General Hospital ( Site 0929), Kobe, Hyōgo
  - Ibaraki Prefectural Central Hospital ( Site 0918), Kasama, Ibaraki
  - University of Tsukuba Hospital ( Site 0910), Tsukuba, Ibaraki
  - Kagawa University Hospital ( Site 0915), Kita-gun, Kagawa-ken
  - St. Marianna University School of Medicine Hospital ( Site 0903), Kawasaki, Kanagawa
  - Kanagawa Cancer Center ( Site 0921), Yokohama, Kanagawa
  - Oita University Hospital ( Site 0930), Yufu, Oita Prefecture
  - Kansai Medical University Hospital ( Site 0931), Hirakata, Osaka
  - Kindai University Hospital ( Site 0917), Sayama, Osaka
  - Osaka University Hospital ( Site 0911), Suita, Osaka
  - Osaka Medical College Hospital ( Site 0925), Takatsuki, Osaka
  - Saitama Cancer Center ( Site 0926), Kitaadachi-gun, Saitama
  - Shizuoka Cancer Center Hospital and Research Institute ( Site 0914), Sunto-gun, Shizuoka
  - Kyorin University Hospital ( Site 0905), Mitaka, Tokyo
  - Chiba University Hospital ( Site 0909), Chiba
  - Chiba Cancer Center ( Site 0900), Chiba
  - National Hospital Organization Kyushu Cancer Center ( Site 0906), Fukuoka
  - Kyushu University Hospital ( Site 0922), Fukuoka
  - Gifu University Hospital ( Site 0920), Gifu
  - Kumamoto University Hospital ( Site 0919), Kumamoto
  - Niigata Cancer Center Hospital ( Site 0924), Niigata
  - Osaka International Cancer Institute ( Site 0923), Osaka
  - Osaka General Medical Center ( Site 0912), Osaka
  - National Cancer Center Hospital ( Site 0907), Tokyo
  - The Cancer Institute Hospital of JFCR ( Site 0904), Tokyo
  - Keio University Hospital ( Site 0927), Tokyo
- Malaysia (3):
  - Beacon International Specialist Centre ( Site 1803), Petaling Jaya, Selangor
  - Hospital Kuala Lumpur ( Site 1805), Kuala Lumpur
  - University Malaya Medical Centre ( Site 1802), Kuala Lumpur
- Peru (3):
  - Instituto Regional de Enfermedades Neoplasicas del Sur IRENSUR ( Site 1702), Arequipa
  - Hospital Nacional Guillermo Almenara Irigoyen ( Site 1701), Lima
  - Instituto Nacional de Enfermedades Neoplasicas ( Site 1705), Lima
- Romania (7):
  - S C Pelican Impex SRL ( Site 2403), Oradea, Bihor County
  - S.C. Radiotherapy Center Cluj S.R.L ( Site 2407), Comuna Floresti, Cluj
  - S.C. Centrul de Oncologie Sf. Nectarie SRL ( Site 2404), Craiova, Dolj
  - S.C.Focus Lab Plus S.R.L ( Site 2401), Bucharest, Sector 2
  - S C Oncocenter Oncologie Medicala S R L ( Site 2405), Timișoara, Timiș County
  - S.C.Gral Medical S.R.L ( Site 2406), Bucharest
  - Spitalul Clinic Judetean De Urgenta Constanta ( Site 2402), Constanța
- Russia (7):
  - SBHCI RCOD of MHC RB ( Site 0407), Ufa, Bashkortostan Republic
  - Leningrad Regional Oncology Center ( Site 0405), Saint Petersburg, Vsevolzhsk District
  - National Medical and Surgical Center n.a. N.I.Pirogov ( Site 0402), Moscow
  - N.N. Blokhin NMRCO ( Site 0401), Moscow
  - Scientific Research Oncology Institute n.a. N.N.Petrov ( Site 0406), Saint Petersburg
  - St Petersburg City Clinical Oncology Dispensary ( Site 0409), Saint Petersburg
  - Tomsk Scientific Research Institute of Oncology ( Site 0403), Tomsk
- South Africa (7):
  - Cancer Care Langenhoven Drive Oncology Centre ( Site 2501), Port Elizabeth, Eastern Cape
  - The Medical Oncology Centre of Rosebank ( Site 2506), Johannesburg, Gauteng
  - WITS Clinical Research CMJAH Clinical Trial Site ( Site 2500), Parktown, Gauteng
  - The Oncology Centre ( Site 2502), Durban, KwaZulu-Natal
  - Cape Town Oncology Trials Pty Ltd ( Site 2508), Cape Town, Western Cape
  - Outeniqua Cancercare Oncology Unit ( Site 2504), George, Western Cape
  - Clinton Oncology Centre ( Site 2505), Alberton
- South Korea (6):
  - National Cancer Center ( Site 1304), Goyang-si, Gyeonggi-do
  - Chonnam National University Hwasun Hospital ( Site 1305), Hwasun Gun, Jeollanam-do
  - Seoul National University Cancer Hospital ( Site 1301), Seoul
  - Severance Hospital Yonsei University Health System ( Site 1302), Seoul
  - Asan Medical Center ( Site 1303), Seoul
  - Samsung Medical Center ( Site 1300), Seoul
- Spain (7):
  - Hosp. Gral. Universitari Germans Trias i Pujol ( Site 0701), Badalona, Barcelona
  - Hospital Universitario Central de Asturias ( Site 0708), Oviedo, Principality of Asturias
  - Hospital Universitari Vall d Hebron ( Site 0702), Barcelona
  - Hospital Universitario Reina Sofia ( Site 0706), Córdoba
  - Hospital Ramon y Cajal ( Site 0703), Madrid
  - Hospital Universitario La Paz ( Site 0700), Madrid
  - Complejo Hospitalario Virgen De La Victoria ( Site 0705), Málaga
- Taiwan (9):
  - Chang Gung Med Foundation. Kaohsiung Branch ( Site 1906), Kaohsiung City
  - Taipei Medical University Shuang Ho Hospital ( Site 1908), New Taipei City
  - China Medical University Hospital ( Site 1904), Taichung
  - Kuang Tien General Hospital ( Site 1909), Taichung
  - National Cheng Kung University Hospital ( Site 1905), Tainan
  - Chi Mei Medical Center Liuying ( Site 1907), Tainan
  - National Taiwan University Hospital ( Site 1900), Taipei
  - Koo Foundation Sun Yat-Sen Cancer Center ( Site 1902), Taipei
  - Chang Gung Medical Foundation. Linkou ( Site 1903), Taoyuan District
- Thailand (5):
  - Bumrungrad International Hospital ( Site 2203), Bangkok
  - Chulalongkorn Hospital ( Site 2201), Bangkok
  - Ramathibodi Hospital. ( Site 2202), Bangkok
  - Phramongkutklao Hospital ( Site 2205), Bangkok
  - Songklanagarind Hospital ( Site 2204), Songkhla
- Turkey (Türkiye) (7):
  - Adana Sehir Hastanesi ( Site 0802), Adana
  - Ankara Sehir Hastanesi ( Site 0808), Ankara
  - Istanbul Medeniyet Universitesi Goztepe EAH ( Site 0807), Istanbul
  - Istanbul Universitesi Cerrahpasa Tip Fakultesi ( Site 0804), Istanbul
  - Marmara Universitesi Pendik Egitim ve Arastirma Hastanesi ( Site 0801), Istanbul
  - Medical Park Izmir Hastanesi ( Site 0800), Izmir
  - Inonu Universitesi Turgut Ozal Tip Merkezi ( Site 0803), Malatya
- United Kingdom (3):
  - Lothian University Hospitals NHS Trust ( Site 1101), Edinburgh, Mid Lothian
  - St Luke's Cancer Centre ( Site 1102), Guildford
  - The Christie NHS Foundation Trust ( Site 1100), Manchester

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Mansoor W, Joo S, Norquist JM, Kato K, Sun JM, Shah MA, Enzinger P, Adenis A, Doi T, Kojima T, Metges JP, Li Z, Kim SB, Cho BC, Sunpaweravong P, Alsina M, Goekkurt E, Suryawanshi S, Shah S, Shen L. Health-related quality-of-life analysis from KEYNOTE-590: pembrolizumab plus chemotherapy versus chemotherapy for advanced esophageal cancer. Oncologist. 2024 Oct 3;29(10):e1324-e1335. doi: 10.1093/oncolo/oyae087. PMID 38815152
- [Derived] Kato K, Kojima T, Hara H, Tsuji A, Yasui H, Muro K, Satoh T, Ogata T, Ishihara R, Goto M, Baba H, Nishina T, Han S, Iwakami K, Yatsuzuka N, Doi T. First-line pembrolizumab plus chemotherapy for advanced/metastatic esophageal cancer: 1-year extended follow-up in the Japanese subgroup of the phase 3 KEYNOTE-590 study. Esophagus. 2024 Jul;21(3):306-318. doi: 10.1007/s10388-024-01053-z. Epub 2024 Apr 12. PMID 38607538
- [Derived] Zhang Y, Li C, Du K, Pengkhun N, Huang Z, Gong M, Li Y, Liu X, Li L, Wang D, Wang C, Chen F, Li J. Comparative analysis of immune checkpoint inhibitors in first-line treatment of esophageal squamous cell carcinoma: a network meta-analysis. Immunotherapy. 2023 Jul;15(10):737-750. doi: 10.2217/imt-2022-0236. Epub 2023 May 4. PMID 37139963
- [Derived] Kojima T, Hara H, Tsuji A, Yasui H, Muro K, Satoh T, Ogata T, Ishihara R, Goto M, Baba H, Nishina T, Han S, Sakata T, Yatsuzuka N, Doi T, Kato K. First-line pembrolizumab + chemotherapy in Japanese patients with advanced/metastatic esophageal cancer from KEYNOTE-590. Esophagus. 2022 Oct;19(4):683-692. doi: 10.1007/s10388-022-00920-x. Epub 2022 Jun 7. PMID 35668304
- [Derived] Zhu Y, Liu K, Ding D, Zhou Y, Peng L. Pembrolizumab Plus Chemotherapy as First-Line Treatment for Advanced Esophageal Cancer: A Cost-Effectiveness Analysis. Adv Ther. 2022 Jun;39(6):2614-2629. doi: 10.1007/s12325-022-02101-9. Epub 2022 Apr 8. PMID 35394255
- [Derived] Sun JM, Shen L, Shah MA, Enzinger P, Adenis A, Doi T, Kojima T, Metges JP, Li Z, Kim SB, Cho BC, Mansoor W, Li SH, Sunpaweravong P, Maqueda MA, Goekkurt E, Hara H, Antunes L, Fountzilas C, Tsuji A, Oliden VC, Liu Q, Shah S, Bhagia P, Kato K; KEYNOTE-590 Investigators. Pembrolizumab plus chemotherapy versus chemotherapy alone for first-line treatment of advanced oesophageal cancer (KEYNOTE-590): a randomised, placebo-controlled, phase 3 study. Lancet. 2021 Aug 28;398(10302):759-771. doi: 10.1016/S0140-6736(21)01234-4. PMID 34454674
- [Derived] Kato K, Shah MA, Enzinger P, Bennouna J, Shen L, Adenis A, Sun JM, Cho BC, Ozguroglu M, Kojima T, Kostorov V, Hierro C, Zhu Y, McLean LA, Shah S, Doi T. KEYNOTE-590: Phase III study of first-line chemotherapy with or without pembrolizumab for advanced esophageal cancer. Future Oncol. 2019 Apr;15(10):1057-1066. doi: 10.2217/fon-2018-0609. Epub 2019 Feb 8. PMID 30735435
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26081&tenant=MT_MSD_9011

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 749 participants were randomized 1:1 to receive either pembrolizumab plus standard of care (SOC) chemotherapy, or placebo plus SOC chemotherapy.
Groups:
- Pembrolizumab + SOC: Participants received pembrolizumab 200 mg intravenously (IV) every 3 weeks (Q3W) plus standard of care (SOC) chemotherapy with cisplatin 80 mg/m^2 IV Q3W and 5-fluorouracil (5-FU) 800 mg/m^2/day continuous IV infusion on Days 1 to 5 (120 hours) Q3W. All treatments were administered on an outpatient basis beginning on Day 1 of each 3-week dosing cycle.
- Placebo + SOC: Participants received placebo to pembrolizumab (saline) IV Q3W plus SOC chemotherapy with cisplatin 80 mg/m^2 IV Q3W and 5-FU 800 mg/m^2/day continuous IV infusion on Days 1 to 5 (120 hours) Q3W. All treatments were administered on an outpatient basis beginning on Day 1 of each 3-week dosing cycle.
Period: Overall Study
Arm/Group | Pembrolizumab + SOC | Placebo + SOC
Started | 373 | 376
Treated | 370 | 370
Completed | 0 | 0
Not Completed | 373 | 376
Not completed — Death | 325 | 361
Not completed — Physician Decision | 1 | 0
Not completed — Sponsor Decision | 40 | 12
Not completed — Withdrawal by Subject | 7 | 3

BASELINE CHARACTERISTICS:
Groups:
- Pembrolizumab + SOC: Participants received pembrolizumab 200 mg IV Q3W plus SOC chemotherapy with cisplatin 80 mg/m^2 IV Q3W and 5-FU 800 mg/m^2/day continuous IV infusion on Days 1 to 5 (120 hours) Q3W. All treatments were administered on an outpatient basis beginning on Day 1 of each 3-week dosing cycle.
- Total: Total of all reporting groups
Arm/Group | Pembrolizumab + SOC | Placebo + SOC | Total
Number analyzed (Participants) | 373 | 376 | 749
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.8 (9.8) | 62.0 (9.2) | 62.4 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67 | 57 | 124
  Male | 306 | 319 | 625
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 42 | 57 | 99
  Not Hispanic or Latino | 315 | 296 | 611
  Unknown or Not Reported | 16 | 23 | 39
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 9 | 12 | 21
  Asian | 201 | 199 | 400
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 2 | 7
  White | 139 | 139 | 278
  More than one race | 5 | 9 | 14
  Unknown or Not Reported | 14 | 15 | 29
Geographic Region [Count of Participants; unit: Participants] — Participants were stratified according to Geographic Region of enrolling site (Asia versus Rest of World)
  Participants
    Asia | 196 | 197 | 393
    Rest of World | 177 | 179 | 356
Histology [Count of Participants; unit: Participants] — Participants were stratified according to baseline Histology (adenocarcinoma versus squamous cell carcinoma)
  Participants
    Adenocarcinoma | 99 | 102 | 201
    Squamous Cell Carcinoma | 274 | 274 | 548
Eastern Cooperative Group Performance Status (ECOG PS) [Count of Participants; unit: Participants] — ECOG PS 0 = Fully active, able to carry on all pre-disease performance without restriction), ECOG PS 1 = Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, ECOG PS 2 = Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours. Participants were stratified according to baseline ECOG PS (0 versus 1).
  Participants
    ECOG PS 0 | 149 | 150 | 299
    ECOG PS 1 | 223 | 225 | 448
    ECOG PS 2 | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS) in Participants With Esophageal Squamous Cell Carcinoma (ESCC) Whose Tumors Are Programmed Cell Death-Ligand 1 (PD-L1) Biomarker-Positive (Combined Positive Score [CPS] ≥10)
Description: Overall survival was defined as the time from randomization to death due to any cause. Participants without documented death at the time of the final analysis were censored at the date of the last follow-up. Per protocol, OS is reported here for all participants of the Intent-To-Treat (ITT) population (all randomized) who had ESCC and who were PD-L1 CPS ≥10.
Time Frame: Up to approximately 34 months
Population: All randomized participants (ITT population) with ESCC and PD-L1 CPS ≥10 were analyzed.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + SOC | Placebo + SOC
Number analyzed (Participants) | 143 | 143
Months | 13.9 [11.1 to 17.7] | 8.8 [7.8 to 10.5]
Statistical Analysis 1: Comparison: Pembrolizumab + SOC vs Placebo + SOC; OS in ESCC PD-L1 CPS ≥10 participants of the pembrolizumab + SOC arm was compared to OS in ESCC PD-L1 CPS ≥10 participants of the placebo + SOC arm based on a Cox regression model with Efron's method of tie handling with treatment as a covariate stratified by geographic region (Asia versus Rest of the World) and ECOG performance status (0 versus 1); Test type: Superiority; p < 0.0001, Stratified Log-Rank; Hazard Ratio (HR) = 0.57, 95% CI 2-sided [0.43 to 0.75]

2. Primary Outcome: OS in Participants With ESCC
Description: Overall survival was defined as the time from randomization to death due to any cause. Participants without documented death at the time of the final analysis were censored at the date of the last follow-up. Per protocol, OS is reported here for all participants of the ITT population (all randomized) who had ESCC.
Time Frame: Up to approximately 34 months
Population: All randomized participants (ITT population) with ESCC were analyzed.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + SOC | Placebo + SOC
Number analyzed (Participants) | 274 | 274
Months | 12.6 [10.2 to 14.3] | 9.8 [8.6 to 11.1]
Statistical Analysis 1: Comparison: Pembrolizumab + SOC vs Placebo + SOC; OS in ESCC participants of the pembrolizumab + SOC arm was compared to OS in ESCC participants of the placebo + SOC arm based on a Cox regression model with Efron's method of tie handling with treatment as a covariate stratified by geographic region (Asia versus Rest of the World) and ECOG performance status (0 versus 1); Test type: Superiority; p = 0.0006, Stratified Log-Rank; Hazard Ratio (HR) = 0.72, 95% CI 2-sided [0.60 to 0.88]

3. Primary Outcome: OS in Participants Whose Tumors Are PD-L1 Biomarker-Positive (CPS ≥10)
Description: Overall survival was defined as the time from randomization to death due to any cause. Participants without documented death at the time of the final analysis were censored at the date of the last follow-up. Per protocol, OS is reported here for all participants of the ITT population (all randomized) who were PD-L1 CPS ≥10.
Time Frame: Up to approximately 34 months
Population: All randomized participants (ITT population) who were PD-L1 CPS ≥10 were analyzed.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + SOC | Placebo + SOC
Number analyzed (Participants) | 186 | 197
Months | 13.5 [11.1 to 15.6] | 9.4 [8.0 to 10.7]
Statistical Analysis 1: Comparison: Pembrolizumab + SOC vs Placebo + SOC; OS in PD-L1 CPS ≥10 participants of the pembrolizumab + SOC arm was compared to OS in PD-L1 CPS ≥10 participants of the placebo + SOC arm based on a Cox regression model with Efron's method of tie handling with treatment as a covariate stratified by geographic region (Asia versus Rest of the World) and tumor histology (Adenocarcinoma versus Squamous Cell Carcinoma); Test type: Superiority; p < 0.0001, Stratified Log-Rank; Hazard Ratio (HR) = 0.62, 95% CI 2-sided [0.49 to 0.78]

4. Primary Outcome: OS in All Participants
Description: Overall survival was defined as the time from randomization to death due to any cause. Participants without documented death at the time of the final analysis were censored at the date of the last follow-up. Per protocol, OS is reported here for all participants of the ITT population (all randomized).
Time Frame: Up to approximately 34 months
Population: All randomized participants (ITT population) were analyzed.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + SOC | Placebo + SOC
Number analyzed (Participants) | 373 | 376
Months | 12.4 [10.5 to 14.0] | 9.8 [8.8 to 10.8]
Statistical Analysis 1: Comparison: Pembrolizumab + SOC vs Placebo + SOC; OS in all participants of the pembrolizumab + SOC arm was compared to OS in all participants of the placebo + SOC arm based on a Cox regression model with Efron's method of tie handling with treatment as a covariate stratified by geographic region (Asia versus Rest of the World), tumor histology (Adenocarcinoma versus Squamous Cell Carcinoma), and ECOG performance status (0 versus 1); Test type: Superiority; p < 0.0001, Stratified Log-Rank; Hazard Ratio (HR) = 0.73, 95% CI 2-sided [0.62 to 0.86]

5. Primary Outcome: Progression-free Survival (PFS) Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) As Assessed By Investigator in Participants With ESCC
Description: PFS was defined as the time from randomization to the first documented progressive disease (PD) per RECIST 1.1 as assessed by the investigator, or death due to any cause, whichever occurred first. Per RECIST 1.1, PD was defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum had to demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions was also considered PD. The sponsor allowed a maximum of 10 target lesions in total and 5 per organ on this study. Per protocol, PFS is reported here for all participants of the ITT population (all randomized) who had ESCC.
Time Frame: Up to approximately 34 months
Population: All randomized participants (ITT population) with ESCC were analyzed.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + SOC | Placebo + SOC
Number analyzed (Participants) | 274 | 274
Months | 6.3 [6.2 to 6.9] | 5.8 [5.0 to 6.1]
Statistical Analysis 1: Comparison: Pembrolizumab + SOC vs Placebo + SOC; PFS in ESCC participants of the pembrolizumab + SOC arm was compared to PFS in ESCC participants of the placebo + SOC arm based on a Cox regression model with Efron's method of tie handling with treatment as a covariate stratified by geographic region (Asia versus Rest of the World) and ECOG performance status (0 versus 1); Test type: Superiority; p < 0.0001, Stratified Log-Rank; Hazard Ratio (HR) = 0.65, 95% CI 2-sided [0.54 to 0.78]

6. Primary Outcome: PFS Per RECIST 1.1 As Assessed By Investigator in Participants Whose Tumors Are PD-L1 Biomarker-Positive (CPS ≥10)
Description: PFS was defined as the time from randomization to the first documented progressive disease (PD) per RECIST 1.1 as assessed by the investigator, or death due to any cause, whichever occurred first. Per RECIST 1.1, PD was defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum had to demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions was also considered PD. The sponsor allowed a maximum of 10 target lesions in total and 5 per organ on this study. Per protocol, PFS is reported here for all participants of the ITT population (all randomized) who were PD-L1 CPS ≥10.
Time Frame: Up to approximately 34 months
Population: All randomized participants (ITT population) who were PD-L1 CPS ≥10 were analyzed.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + SOC | Placebo + SOC
Number analyzed (Participants) | 186 | 197
Months | 7.5 [6.2 to 8.2] | 5.5 [4.3 to 6.0]
Statistical Analysis 1: Comparison: Pembrolizumab + SOC vs Placebo + SOC; PFS in PD-L1 CPS ≥10 participants of the pembrolizumab + SOC arm was compared to PFS in PD-L1 CPS ≥10 participants of the placebo + SOC arm based on a Cox regression model with Efron's method of tie handling with treatment as a covariate stratified by geographic region (Asia versus Rest of the World) and tumor histology (Adenocarcinoma versus Squamous Cell Carcinoma); Test type: Superiority; p < 0.0001, Stratified Log-Rank; Hazard Ratio (HR) = 0.51, 95% CI 2-sided [0.41 to 0.65]

7. Primary Outcome: PFS Per RECIST 1.1 As Assessed By Investigator in All Participants
Description: PFS was defined as the time from randomization to the first documented progressive disease (PD) per RECIST 1.1 as assessed by the investigator, or death due to any cause, whichever occurred first. Per RECIST 1.1, PD was defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum had to demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions was also considered PD. The sponsor allowed a maximum of 10 target lesions in total and 5 per organ on this study. Per protocol, PFS is reported here for all participants of the ITT population (all randomized).
Time Frame: Up to approximately 34 months
Population: All randomized participants (ITT population) were analyzed.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + SOC | Placebo + SOC
Number analyzed (Participants) | 373 | 376
Months | 6.3 [6.2 to 6.9] | 5.8 [5.0 to 6.0]
Statistical Analysis 1: Comparison: Pembrolizumab + SOC vs Placebo + SOC; PFS in all participants of the pembrolizumab + SOC arm was compared to PFS in all participants of the placebo + SOC arm based on a Cox regression model with Efron's method of tie handling with treatment as a covariate stratified by geographic region (Asia versus Rest of the World), tumor histology (Adenocarcinoma versus Squamous Cell Carcinoma), and ECOG performance status (0 versus 1); Test type: Superiority; p < 0.0001, Stratified Log-Rank; Hazard Ratio (HR) = 0.65, 95% CI 2-sided [0.55 to 0.76]

8. Secondary Outcome: Objective Response Rate (ORR) Per RECIST 1.1 As Assessed By Investigator in All Participants
Description: ORR was defined as the percentage of participants in the analysis population who had a Complete Response (CR: disappearance of all target lesions) or a Partial Response (PR: ≥30% decrease in the sum of diameters of target lesions) per RECIST 1.1. as assessed by the investigator. The sponsor allowed a maximum of 10 target lesions in total and 5 per organ on this study. Per protocol, the percentage of participants who experienced CR or PR is reported here as the ORR for all participants of the ITT population (all randomized).
Time Frame: Up to approximately 34 months
Population: All randomized participants (ITT population) were analyzed.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Pembrolizumab + SOC | Placebo + SOC
Number analyzed (Participants) | 373 | 376
Percentage of Participants | 45.0 [39.9 to 50.2] | 29.3 [24.7 to 34.1]
Statistical Analysis 1: Comparison: Pembrolizumab + SOC vs Placebo + SOC; ORR in all participants of the pembrolizumab + SOC arm was compared to ORR in all participants of the placebo + SOC arm based on the Miettinen & Nurminen method stratified by geographic region (Asia versus Rest of the World), tumor histology (Adenocarcinoma versus Squamous Cell Carcinoma), and ECOG performance status (0 versus 1); Test type: Superiority; p < 0.0001, One-sided p-value; Difference in Percentage = 15.8, 95% CI 2-sided [9.0 to 22.5]

9. Secondary Outcome: ORR Per RECIST 1.1 As Assessed By Investigator in Participants With ESCC Whose Tumors Are PD-L1 Biomarker-Positive (CPS ≥10)
Description: ORR was defined as the percentage of participants in the analysis population who had a Complete Response (CR: disappearance of all target lesions) or a Partial Response (PR: ≥30% decrease in the sum of diameters of target lesions) per RECIST 1.1. as assessed by the investigator. The sponsor allowed a maximum of 10 target lesions in total and 5 per organ on this study. Per protocol, the percentage of participants who experienced CR or PR is reported here as the ORR for all participants of the ITT population (all randomized) who had ESCC and who were PD-L1 CPS ≥10.
Time Frame: Up to approximately 34 months
Population: All randomized participants (ITT population) with ESCC and PD-L1 CPS ≥10 were analyzed.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Pembrolizumab + SOC | Placebo + SOC
Number analyzed (Participants) | 143 | 143
Percentage of Participants | 51.0 [42.6 to 59.5] | 28.0 [20.8 to 36.1]
Statistical Analysis 1: Comparison: Pembrolizumab + SOC vs Placebo + SOC; ORR in ESCC PD-L1 CPS ≥10 participants of the pembrolizumab + SOC arm was compared to ORR in ESCC PD-L1 CPS ≥10 participants of the placebo + SOC arm based on the Miettinen & Nurminen method stratified by geographic region (Asia versus Rest of the World) and ECOG performance status (0 versus 1); Test type: Other; p < 0.0001, One-sided p-value; Difference in Percentage = 22.8, 95% CI 2-sided [11.6 to 33.4]

10. Secondary Outcome: ORR Per RECIST 1.1 As Assessed By Investigator in Participants With ESCC
Description: ORR was defined as the percentage of participants in the analysis population who had a Complete Response (CR: disappearance of all target lesions) or a Partial Response (PR: ≥30% decrease in the sum of diameters of target lesions) per RECIST 1.1. as assessed by the investigator. The sponsor allowed a maximum of 10 target lesions in total and 5 per organ on this study. Per protocol, the percentage of participants who experienced CR or PR is reported here as the ORR for all participants of the ITT population (all randomized) who had ESCC.
Time Frame: Up to approximately 34 months
Population: All randomized participants (ITT population) with ESCC were analyzed.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Pembrolizumab + SOC | Placebo + SOC
Number analyzed (Participants) | 274 | 274
Percentage of Participants | 43.8 [37.8 to 49.9] | 31.0 [25.6 to 36.9]
Statistical Analysis 1: Comparison: Pembrolizumab + SOC vs Placebo + SOC; ORR in ESCC participants of the pembrolizumab + SOC arm was compared to ORR in ESCC participants of the placebo + SOC arm based on the Miettinen & Nurminen method stratified by geographic region (Asia versus Rest of the World) and ECOG performance status (0 versus 1); Test type: Other; p = 0.0009, One-sided p-value; Difference in Percentage = 12.8, 95% CI 2-sided [4.7 to 20.7]

11. Secondary Outcome: ORR Per RECIST 1.1 As Assessed By Investigator in Participants Whose Tumors Are PD-L1 Biomarker-Positive (CPS ≥10)
Description: ORR was defined as the percentage of participants in the analysis population who had a Complete Response (CR: disappearance of all target lesions) or a Partial Response (PR: ≥30% decrease in the sum of diameters of target lesions) per RECIST 1.1. as assessed by the investigator. The sponsor allowed a maximum of 10 target lesions in total and 5 per organ on this study. Per protocol, the percentage of participants who experienced CR or PR is reported here as the ORR for all participants of the ITT population (all randomized) who were PD-L1 CPS ≥10.
Time Frame: Up to approximately 34 months
Population: All randomized participants (ITT population) who were PD-L1 CPS ≥10 were analyzed.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Pembrolizumab + SOC | Placebo + SOC
Number analyzed (Participants) | 186 | 197
Percentage of Participants | 51.1 [43.7 to 58.5] | 26.9 [20.8 to 33.7]
Statistical Analysis 1: Comparison: Pembrolizumab + SOC vs Placebo + SOC; ORR in PD-L1 CPS ≥10 participants of the pembrolizumab + SOC arm was compared to ORR in PD-L1 CPS ≥10 participants of the placebo + SOC arm based on the Miettinen & Nurminen method stratified by geographic region (Asia versus Rest of the World) and tumor histology (Adenocarcinoma versus Squamous Cell Carcinoma); Test type: Other; p < 0.0001, One-sided p-value; Difference in Percentage = 24.0, 95% CI 2-sided [14.3 to 33.2]

12. Secondary Outcome: Duration of Response (DOR) Per RECIST 1.1 As Assessed By Investigator in All Participants
Description: For participants who demonstrated a confirmed CR (disappearance of all target lesions) or PR (at least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1 as assessed by the investigator, DOR was defined as the time from first documented evidence of confirmed CR or PR until PD or death due to any cause, whichever occurred first. DOR for participants who had not progressed or died at the time of analysis was censored at the date of their last tumor assessment. Per RECIST 1.1, PD was defined as at least a 20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum had to demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions was also considered PD. Per protocol, DOR is reported here for all participants of the ITT population (all randomized) who had CR or PR.
Time Frame: Up to approximately 34 months
Population: All randomized participants (ITT population) who demonstrated a confirmed CR or PR were analyzed.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + SOC | Placebo + SOC
Number analyzed (Participants) | 168 | 110
Months | 8.3 [6.4 to 10.4] | 6.0 [4.4 to 6.4]

13. Secondary Outcome: DOR Per RECIST 1.1 As Assessed By Investigator in Participants With ESCC Whose Tumors Are PD-L1 Biomarker-Positive (CPS ≥10)
Description: For participants who demonstrated a confirmed CR (disappearance of all target lesions) or PR (at least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1 as assessed by the investigator, DOR was defined as the time from first documented evidence of confirmed CR or PR until PD or death due to any cause, whichever occurred first. DOR for participants who had not progressed or died at the time of analysis was censored at the date of their last tumor assessment. Per RECIST 1.1, PD was defined as at least a 20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum had to demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions was also considered PD. Per protocol, DOR is reported here for all participants of the ITT population (all randomized) who had CR or PR, and who had ESCC and were PD-L1 CPS ≥10.
Time Frame: Up to approximately 34 months
Population: All randomized participants (ITT population) with ESCC and PD-L1 CPS ≥10 who demonstrated a confirmed CR or PR were analyzed were analyzed.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + SOC | Placebo + SOC
Number analyzed (Participants) | 73 | 40
Months | 10.4 [8.0 to 16.2] | 4.4 [4.1 to 6.2]

14. Secondary Outcome: DOR Per RECIST 1.1 As Assessed By Investigator in Participants With ESCC
Description: For participants who demonstrated a confirmed CR (disappearance of all target lesions) or PR (at least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1 as assessed by the investigator, DOR was defined as the time from first documented evidence of confirmed CR or PR until PD or death due to any cause, whichever occurred first. DOR for participants who had not progressed or died at the time of analysis was censored at the date of their last tumor assessment. Per RECIST 1.1, PD was defined as at least a 20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum had to demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions was also considered PD. Per protocol, DOR is reported here for all participants of the ITT population (all randomized) who had CR or PR, and who had ESCC.
Time Frame: Up to approximately 34 months
Population: All randomized participants (ITT population) with ESCC who demonstrated a confirmed CR or PR were analyzed.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + SOC | Placebo + SOC
Number analyzed (Participants) | 120 | 85
Months | 9.1 [6.6 to 12.3] | 6.1 [4.4 to 6.4]

15. Secondary Outcome: DOR Per RECIST 1.1 As Assessed By Investigator in Participants Whose Tumors Are PD-L1 Biomarker-Positive (CPS ≥10)
Description: For participants who demonstrated a confirmed CR (disappearance of all target lesions) or PR (at least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1 as assessed by the investigator, DOR was defined as the time from first documented evidence of confirmed CR or PR until PD or death due to any cause, whichever occurred first. DOR for participants who had not progressed or died at the time of analysis was censored at the date of their last tumor assessment. Per RECIST 1.1, PD was defined as at least a 20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum had to demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions was also considered PD. Per protocol, DOR is reported here for all participants of the ITT population (all randomized) who had CR or PR, and were PD-L1 CPS ≥10.
Time Frame: Up to approximately 34 months
Population: All randomized participants (ITT population) who were PD-L1 CPS ≥10 and who demonstrated a confirmed CR or PR were analyzed.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + SOC | Placebo + SOC
Number analyzed (Participants) | 95 | 53
Months | 10.4 [6.7 to 14.5] | 5.6 [4.3 to 6.5]

16. Secondary Outcome: Number of Participants With an Adverse Event (AE)
Description: An AE was defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which did not necessarily have to have a causal relationship with this treatment. An AE could therefore be any unfavourable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening of a pre-existing condition that was temporally associated with the use of the Sponsor's product was also an AE. The number of participants that experienced at least one AE was reported for each treatment arm.
Time Frame: Up to approximately 28 months
Population: All randomized participants who received at least one dose of study treatment were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab + SOC | Placebo + SOC
Number analyzed (Participants) | 370 | 370
Participants | 370 | 368

17. Secondary Outcome: Number of Participants Discontinuing Study Treatment Due to an AE
Description: An AE was defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which did not necessarily have to have a causal relationship with this treatment. An AE could therefore be any unfavourable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening of a pre-existing condition that was temporally associated with the use of the Sponsor's product was also an AE. The number of participants that discontinued any study drug due to an AE was reported for each treatment arm.
Time Frame: Up to approximately 27 months
Population: All randomized participants who received at least one dose of study treatment were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab + SOC | Placebo + SOC
Number analyzed (Participants) | 370 | 370
Participants | 90 | 74

18. Secondary Outcome: Change From Baseline To Week 18 in the European Organization for the Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire C30 (QLQ-C30) Global Health Status/Quality of Life (GHS/QoL) Combined Score in All Participants
Description: The EORTC-QLQ-C30 is a 30-item questionnaire developed to assess the quality of life of cancer patients. Participant responses to the Global Health Status (GHS) question "How would you rate your overall health during the past week?" (Item 29) and the Quality of Life (QoL) question "How would you rate your overall quality of life during the past week?" (Item 30) were scored on a 7-point scale (1=Very Poor to 7=Excellent). Using linear transformation, raw scores were standardized so that scores ranged from 0 to 100, with a higher score indicating a better overall outcome. Per protocol, change from baseline to Week 18 in the GHS/QoL combined score was reported by treatment arm as a pre-specified secondary analysis for all participants.
Time Frame: Baseline, Week 18
Population: All randomized participants who received at least one dose of study treatment and completed at least 1 EORTC-QLQ-C30 assessment were analyzed.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a Scale
Arm/Group | Pembrolizumab + SOC | Placebo + SOC
Number analyzed (Participants) | 366 | 363
Score on a Scale | -1.74 [-4.24 to 0.75] | -1.64 [-4.21 to 0.92]
Statistical Analysis 1: Comparison: Pembrolizumab + SOC vs Placebo + SOC; Change from baseline to Week 18 in EORTC-QLQ-C30 GHS/QoL combined score was compared between treatment arms based on a constrained longitudinal data analysis (cLDA) model with the EORTC-QLQ-C30 GHS/QoL scores as the response variable with covariates for treatment by study visit interaction, and stratification factors including geographic region (Asia versus Rest of the World) and tumor histology (Adenocarcinoma versus Squamous Cell Carcinoma) and ECOG performance status (0 versus 1); Test type: Other; p = 0.9530, constrained Longitudinal Data Analysis; Difference in LS Means = -0.10, 95% CI 2-sided [-3.40 to 3.20]

19. Secondary Outcome: Change From Baseline To Week 18 in the EORTC QLQ-C30 GHS/QoL Combined Score in Participants With ESCC Whose Tumors Are PD-L1 Biomarker-Positive (CPS ≥10)
Description: The EORTC-QLQ-C30 is a 30-item questionnaire developed to assess the quality of life of cancer patients. Participant responses to the Global Health Status (GHS) question "How would you rate your overall health during the past week?" (Item 29) and the Quality of Life (QoL) question "How would you rate your overall quality of life during the past week?" (Item 30) were scored on a 7-point scale (1=Very Poor to 7=Excellent). Using linear transformation, raw scores were standardized so that scores ranged from 0 to 100, with a higher score indicating a better overall outcome. Per protocol, change from baseline to Week 18 in the GHS/QoL combined score was reported by treatment arm as a pre-specified secondary analysis for all participants who had ESCC and who were PD-L1 CPS ≥10.
Time Frame: Baseline, Week 18
Population: All randomized participants who received at least one dose of study treatment, completed at least 1 EORTC-QLQ-C30 assessment, who had ESCC, and who were PD-L1 CPS ≥10 were analyzed.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a Scale
Arm/Group | Pembrolizumab + SOC | Placebo + SOC
Number analyzed (Participants) | 142 | 138
Score on a Scale | -2.36 [-6.58 to 1.87] | -0.40 [-4.86 to 4.05]
Statistical Analysis 1: Comparison: Pembrolizumab + SOC vs Placebo + SOC; Change from baseline to Week 18 in EORTC-QLQ-C30 GHS/QoL combined score was compared between treatment arms based on a cLDA model with the EORTC-QLQ-C30 GHS/QoL scores as the response variable with covariates for treatment by study visit interaction, and stratification factors including geographic region (Asia versus Rest of the World) and ECOG performance status (0 versus 1); Test type: Other; p = 0.5053, constrained Longitudinal Data Analysis; Difference in LS Means = -1.95, 95% CI 2-sided [-7.72 to 3.82]

20. Secondary Outcome: Change From Baseline To Week 18 in the EORTC QLQ-C30 GHS/QoL Combined Score in Participants With ESCC
Description: The EORTC-QLQ-C30 is a 30-item questionnaire developed to assess the quality of life of cancer patients. Participant responses to the Global Health Status (GHS) question "How would you rate your overall health during the past week?" (Item 29) and the Quality of Life (QoL) question "How would you rate your overall quality of life during the past week?" (Item 30) were scored on a 7-point scale (1=Very Poor to 7=Excellent). Using linear transformation, raw scores were standardized so that scores ranged from 0 to 100, with a higher score indicating a better overall outcome. Per protocol, change from baseline to Week 18 in the GHS/QoL combined score was reported by treatment arm as a pre-specified secondary analysis for all participants who had ESCC.
Time Frame: Baseline, Week 18
Population: All randomized participants who received at least one dose of study treatment, completed at least 1 EORTC-QLQ-C30 assessment, and who had ESCC were analyzed.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a Scale
Arm/Group | Pembrolizumab + SOC | Placebo + SOC
Number analyzed (Participants) | 270 | 264
Score on a Scale | -2.00 [-4.90 to 0.89] | -1.94 [-4.93 to 1.06]
Statistical Analysis 1: Comparison: Pembrolizumab + SOC vs Placebo + SOC; [analysis description as in outcome 19, analysis 1]; Test type: Other; p = 0.9742, constrained Longitudinal Data Analysis; Difference in LS Means = -0.06, 95% CI 2-sided [-3.93 to 3.81]

21. Secondary Outcome: Change From Baseline To Week 18 in the EORTC QLQ-C30 GHS/QoL Combined Score in Participants Whose Tumors Are PD-L1 Biomarker-Positive (CPS ≥10)
Description: The EORTC-QLQ-C30 is a 30-item questionnaire developed to assess the quality of life of cancer patients. Participant responses to the Global Health Status (GHS) question "How would you rate your overall health during the past week?" (Item 29) and the Quality of Life (QoL) question "How would you rate your overall quality of life during the past week?" (Item 30) were scored on a 7-point scale (1=Very Poor to 7=Excellent). Using linear transformation, raw scores were standardized so that scores ranged from 0 to 100, with a higher score indicating a better overall outcome. Per protocol, change from baseline to Week 18 in the GHS/QoL combined score was reported by treatment arm as a pre-specified secondary analysis for all participants who were PD-L1 CPS ≥10.
Time Frame: Baseline, Week 18
Population: All randomized participants who received at least one dose of study treatment, completed at least 1 EORTC-QLQ-C30 assessment, and who were PD-L1 CPS ≥10 were analyzed.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a Scale
Arm/Group | Pembrolizumab + SOC | Placebo + SOC
Number analyzed (Participants) | 184 | 191
Score on a Scale | -1.73 [-5.50 to 2.04] | 0.04 [-3.77 to 3.85]
Statistical Analysis 1: Comparison: Pembrolizumab + SOC vs Placebo + SOC; Change from baseline to Week 18 in EORTC-QLQ-C30 GHS/QoL combined score was compared between treatment arms based on a cLDA model with the EORTC-QLQ-C30 GHS/QoL scores as the response variable with covariates for treatment by study visit interaction, and stratification factors including geographic region (Asia versus Rest of the World) and tumor histology (Adenocarcinoma versus Squamous Cell Carcinoma); Test type: Other; p = 0.4810, constrained Longitudinal Data Analysis; Difference in LS Means = -1.77, 95% CI 2-sided [-6.71 to 3.17]

22. Secondary Outcome: Change From Baseline in the EORTC Quality Of Life Questionnaire Oesophageal Module (QLQ-OES18) Subscale Scores in All Participants
Description: The EORTC QLQ-OES18 is a disease-specific questionnaire developed and validated to address measurements specific to esophageal cancer and contains 18 items assessing symptoms of dysphagia, pain, reflux symptoms, eating restrictions, anxiety, dry mouth, taste, body image, and hair loss. For the purposes of this study, the Dysphagia subscale (three items), Pain subscale (three items), and Reflux subscale (two items) were evaluated. All subscale items were scored using a four-point Likert scale with the following response choices: 1=not at all, 2=a little, 3=quite a bit, 4=very much. Raw scores for the subscales were standardized into a range of 0 to 100 by linear transformation, with higher symptom scores represent a higher ("worse") level of symptoms. Per protocol, change from baseline to Week 18 in the Dysphagia, Pain, and Reflux subscales was reported for all participants in each treatment arm. Negative changes from baseline indicate a decrease in symptom severity.
Time Frame: Baseline, Week 18
Population: All randomized participants who received at least one dose of study treatment and completed at least 1 EORTC QLQ-OES18 assessment were analyzed.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a Scale
Arm/Group | Pembrolizumab + SOC | Placebo + SOC
Number analyzed (Participants) | 366 | 359
Score on a Scale
  Dysphagia subscale | -3.18 [-7.19 to 0.82] | 2.36 [-1.77 to 6.49]
  Pain subscale | -4.78 [-7.01 to -2.56] | -1.85 [-4.14 to 0.45]
  Reflux subscale | -0.22 [-2.81 to 2.36] | 0.71 [-1.96 to 3.38]
Statistical Analysis 1: Comparison: Pembrolizumab + SOC vs Placebo + SOC; DYSPHAGIA: Change from baseline to Week 18 in EORTC QLQ-OES18 Dysphagia subscale was compared between treatment arms based on a cLDA model with EORTC QLQ-OES18 scores as the response variable with covariates for treatment by study visit interaction, and stratification factors including geographic region (Asia versus Rest of the World) and tumor histology (Adenocarcinoma versus Squamous Cell Carcinoma) and ECOG performance status (0 versus 1); Test type: Other; p = 0.0436, constrained Longitudinal Data Analysis; Difference in LS Means = -5.54, 95% CI 2-sided [-10.93 to -0.16]
Statistical Analysis 2: Comparison: Pembrolizumab + SOC vs Placebo + SOC; PAIN: Change from baseline to Week 18 in EORTC QLQ-OES18 Pain subscale was compared between treatment arms based on a cLDA model with EORTC QLQ-OES18 scores as the response variable with covariates for treatment by study visit interaction, and stratification factors including geographic region (Asia versus Rest of the World) and tumor histology (Adenocarcinoma versus Squamous Cell Carcinoma) and ECOG performance status (0 versus 1); Test type: Other; p = 0.0487, constrained Longitudinal Data Analysis; Difference in LS Means = -2.94, 95% CI 2-sided [-5.86 to -0.02]
Statistical Analysis 3: Comparison: Pembrolizumab + SOC vs Placebo + SOC; REFLUX: Change from baseline to Week 18 in EORTC QLQ-OES18 Reflux subscale was compared between treatment arms based on a cLDA model with EORTC QLQ-OES18 scores as the response variable with covariates for treatment by study visit interaction, and stratification factors including geographic region (Asia versus Rest of the World) and tumor histology (Adenocarcinoma versus Squamous Cell Carcinoma) and ECOG performance status (0 versus 1); Test type: Other; p = 0.5932, constrained Longitudinal Data Analysis; Difference in LS Means = -0.93, 95% CI 2-sided [-4.36 to 2.49]

23. Secondary Outcome: Change From Baseline in the EORTC QLQ-OES18 Subscale Scores in Participants With ESCC Whose Tumors Are PD-L1 Biomarker-Positive (CPS ≥10)
Description: The EORTC QLQ-OES18 is a disease-specific questionnaire developed and validated to address measurements specific to esophageal cancer and contains 18 items assessing symptoms of dysphagia, pain, reflux symptoms, eating restrictions, anxiety, dry mouth, taste, body image, and hair loss. For the purposes of this study, the Dysphagia subscale (three items), Pain subscale (three items), and Reflux subscale (two items) were evaluated. All subscale items were scored using a four-point Likert scale with the following response choices: 1=not at all, 2=a little, 3=quite a bit, 4=very much. Raw scores for the subscales were standardized into a range of 0 to 100 by linear transformation, with higher symptom scores representing a higher ("worse") level of symptoms. Change from baseline to Week 18 in the Dysphagia, Pain, and Reflux subscales was reported for participants with ESCC who were PD-L1 CPS≥10 in each treatment arm. Negative changes from baseline indicate a decrease in symptom severity.
Time Frame: Baseline, Week 18
Population: All randomized participants who received at least one dose of study treatment, completed at least 1 EORTC QLQ-OES18 assessment, and with ESCC and PD-L1 CPS ≥10 were analyzed.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a Scale
Arm/Group | Pembrolizumab + SOC | Placebo + SOC
Number analyzed (Participants) | 142 | 135
Score on a Scale
  Dysphagia subscale | -5.11 [-11.51 to 1.30] | 3.57 [-3.22 to 10.36]
  Pain subscale | -2.55 [-6.11 to 1.01] | -0.42 [-4.20 to 3.36]
  Reflux subscale | -0.16 [-4.43 to 4.11] | 4.94 [0.43 to 9.46]
Statistical Analysis 1: Comparison: Pembrolizumab + SOC vs Placebo + SOC; DYSPHAGIA: Change from baseline to Week 18 in EORTC QLQ-OES18 Dysphagia subscale was compared between treatment arms based on a cLDA model with EORTC QLQ-OES18 scores as the response variable with covariates for treatment by study visit interaction, and stratification factors including geographic region (Asia versus Rest of the World) and ECOG performance status (0 versus 1); Test type: Other; p = 0.0564, constrained Longitudinal Data Analysis; Difference in LS Means = -8.68, 95% CI 2-sided [-17.59 to 0.24]
Statistical Analysis 2: Comparison: Pembrolizumab + SOC vs Placebo + SOC; PAIN: Change from baseline to Week 18 in EORTC QLQ-OES18 Pain subscale was compared between treatment arms based on a cLDA model with EORTC QLQ-OES18 scores as the response variable with covariates for treatment by study visit interaction, and stratification factors including geographic region (Asia versus Rest of the World) and ECOG performance status (0 versus 1); Test type: Other; p = 0.3813, constrained Longitudinal Data Analysis; Difference in LS Means = -2.13, 95% CI 2-sided [-6.93 to 2.66]
Statistical Analysis 3: Comparison: Pembrolizumab + SOC vs Placebo + SOC; REFLUX: Change from baseline to Week 18 in EORTC QLQ-OES18 Reflux subscale was compared between treatment arms based on a cLDA model with EORTC QLQ-OES18 scores as the response variable with covariates for treatment by study visit interaction, and stratification factors including geographic region (Asia versus Rest of the World) and ECOG performance status (0 versus 1); Test type: Other; p = 0.0816, constrained Longitudinal Data Analysis; Difference in LS Means = -5.11, 95% CI 2-sided [-10.86 to 0.65]

24. Secondary Outcome: Change From Baseline in the EORTC QLQ-OES18 Subscale Scores in Participants With ESCC
Description: The EORTC QLQ-OES18 is a disease-specific questionnaire developed and validated to address measurements specific to esophageal cancer and contains 18 items assessing symptoms of dysphagia, pain, reflux symptoms, eating restrictions, anxiety, dry mouth, taste, body image, and hair loss. For the purposes of this study, the Dysphagia subscale (three items), Pain subscale (three items), and Reflux subscale (two items) were evaluated. All subscale items were scored using a four-point Likert scale with the following response choices: 1=not at all, 2=a little, 3=quite a bit, 4=very much. Raw scores for the subscales were standardized into a range of 0 to 100 by linear transformation, with higher symptom scores representing a higher ("worse") level of symptoms. Change from baseline to Week 18 in the Dysphagia, Pain, and Reflux subscales was reported for participants with ESCC in each treatment arm. Negative changes from baseline indicate a decrease in symptom severity.
Time Frame: Baseline, Week 18
Population: All randomized participants who received at least one dose of study treatment, completed at least 1 EORTC QLQ-OES18 assessment, and with ESCC were analyzed.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a Scale
Arm/Group | Pembrolizumab + SOC | Placebo + SOC
Number analyzed (Participants) | 270 | 261
Score on a Scale
  Dysphagia subscale | -1.18 [-5.82 to 3.47] | 3.32 [-1.50 to 8.13]
  Pain subscale | -4.03 [-6.64 to -1.43] | -2.33 [-5.02 to 0.37]
  Reflux subscale | -0.40 [-3.39 to 2.59] | 1.09 [-2.01 to 4.19]
Statistical Analysis 1: Comparison: Pembrolizumab + SOC vs Placebo + SOC; [analysis description as in outcome 23, analysis 1]; Test type: Other; p = 0.1632, constrained Longitudinal Data Analysis; Difference in LS Means = -4.49, 95% CI 2-sided [-10.81 to 1.83]
Statistical Analysis 2: Comparison: Pembrolizumab + SOC vs Placebo + SOC; [analysis description as in outcome 23, analysis 2]; Test type: Other; p = 0.3259, constrained Longitudinal Data Analysis; Difference in LS Means = -1.71, 95% CI 2-sided [-5.12 to 1.71]
Statistical Analysis 3: Comparison: Pembrolizumab + SOC vs Placebo + SOC; [analysis description as in outcome 23, analysis 3]; Test type: Other; p = 0.4598, constrained Longitudinal Data Analysis; Difference in LS Means = -1.50, 95% CI 2-sided [-5.47 to 2.48]

25. Secondary Outcome: Change From Baseline in the EORTC QLQ-OES18 Subscale Scores in Participants Whose Tumors Are PD-L1 Biomarker-Positive (CPS ≥10)
Description: The EORTC QLQ-OES18 is a disease-specific questionnaire developed and validated to address measurements specific to esophageal cancer and contains 18 items assessing symptoms of dysphagia, pain, reflux symptoms, eating restrictions, anxiety, dry mouth, taste, body image, and hair loss. For the purposes of this study, the Dysphagia subscale (three items), Pain subscale (three items), and Reflux subscale (two items) were evaluated. All subscale items were scored using a four-point Likert scale with the following response choices: 1=not at all, 2=a little, 3=quite a bit, 4=very much. Raw scores for the subscales were standardized into a range of 0 to 100 by linear transformation, with higher symptom scores representing a higher ("worse") level of symptoms. Change from baseline to Week 18 in the Dysphagia, Pain, and Reflux subscales was reported for participants who were PD-L1 CPS≥10 in each treatment arm. Negative changes from baseline indicate a decrease in symptom severity.
Time Frame: Baseline, Week 18
Population: All randomized participants who received at least one dose of study treatment, completed at least 1 EORTC QLQ-OES18 assessment, and with PD-L1 CPS ≥10 were analyzed.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a Scale
Arm/Group | Pembrolizumab + SOC | Placebo + SOC
Number analyzed (Participants) | 184 | 187
Score on a Scale
  Dysphagia subscale | -7.18 [-12.76 to -1.60] | 1.02 [-4.66 to 6.70]
  Pain subscale | -3.51 [-6.69 to -0.33] | 0.07 [-3.18 to 3.31]
  Reflux subscale | -0.52 [-4.17 to 3.14] | 4.25 [0.52 to 7.97]
Statistical Analysis 1: Comparison: Pembrolizumab + SOC vs Placebo + SOC; DYSPHAGIA: Change from baseline to Week 18 in EORTC QLQ-OES18 Dysphagia subscale was compared between treatment arms based on a cLDA model with EORTC QLQ-OES18 scores as the response variable with covariates for treatment by study visit interaction, and stratification factors including geographic region (Asia versus Rest of the World) and tumor histology (Adenocarcinoma versus Squamous Cell Carcinoma); Test type: Other; p = 0.0317, constrained Longitudinal Data Analysis; Difference in LS Means = -8.20, 95% CI 2-sided [-15.67 to -0.73]
Statistical Analysis 2: Comparison: Pembrolizumab + SOC vs Placebo + SOC; PAIN: Change from baseline to Week 18 in EORTC QLQ-OES18 Pain subscale was compared between treatment arms based on a cLDA model with EORTC QLQ-OES18 scores as the response variable with covariates for treatment by study visit interaction, and stratification factors including geographic region (Asia versus Rest of the World) and tumor histology (Adenocarcinoma versus Squamous Cell Carcinoma); Test type: Other; p = 0.0945, constrained Longitudinal Data Analysis; Difference in LS Means = -3.57, 95% CI 2-sided [-7.77 to 0.62]
Statistical Analysis 3: Comparison: Pembrolizumab + SOC vs Placebo + SOC; REFLUX: Change from baseline to Week 18 in EORTC QLQ-OES18 Reflux subscale was compared between treatment arms based on a cLDA model with EORTC QLQ-OES18 scores as the response variable with covariates for treatment by study visit interaction, and stratification factors including geographic region (Asia versus Rest of the World) and tumor histology (Adenocarcinoma versus Squamous Cell Carcinoma); Test type: Other; p = 0.0555, constrained Longitudinal Data Analysis; Difference in LS Means = -4.76, 95% CI 2-sided [-9.64 to 0.11]

ADVERSE EVENTS:
Time Frame: Up to approximately 70 months
Description: All-Cause Mortality table includes all randomized participants, Serious and Other AE tables include all treated participants. Per protocol, disease progression of cancer on study was not considered an AE unless considered related to study drug. Thus, MedDRA preferred terms "Neoplasm progression", "Malignant neoplasm progression" and "Disease progression" not related to study drug were excluded as AEs.
Groups:
- Placebo + SOC: Participants received placebo to pembrolizumab (saline) IV Q3W along with SOC chemotherapy with cisplatin 80 mg/m^2 IV Q3W and 5-FU 800 mg/m^2/day continuous IV infusion on Days 1 to 5 (120 hours) Q3W. All treatments were administered on an outpatient basis beginning on Day 1 of each 3-week dosing cycle.
Arm/Group | Pembrolizumab + SOC | Placebo + SOC
All-Cause Mortality (participants affected / at risk) | 331/373 | 363/376
Serious Adverse Events (participants affected / at risk) | 207/370 | 204/370
Other Adverse Events (participants affected / at risk) | 367/370 | 364/370
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab + SOC (N=370) | Placebo + SOC (N=370)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 10 (10)
Febrile neutropenia (Blood and lymphatic system disorders) | 9 (9) | 13 (13)
Immune thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 5 (5) | 3 (3)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 3 (3)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 2 (2) | 0 (0)
Angina unstable (Cardiac disorders) | 2 (2) | 0 (0)
Arteriospasm coronary (Cardiac disorders) | 1 (1) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 2 (2)
Cardiac failure (Cardiac disorders) | 2 (2) | 2 (2)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1)
Pericarditis (Cardiac disorders) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Tracheo-oesophageal fistula (Congenital, familial and genetic disorders) | 3 (3) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 0 (0)
Graves' disease (Endocrine disorders) | 1 (1) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Hypophysitis (Endocrine disorders) | 1 (1) | 0 (0)
Hypopituitarism (Endocrine disorders) | 1 (1) | 0 (0)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 1 (1) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (4) | 0 (0)
Autoimmune colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 4 (5) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diaphragmatic hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 7 (7) | 5 (5)
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Duodenitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 17 (20) | 13 (13)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Enterocutaneous fistula (Gastrointestinal disorders) | 0 (0) | 1 (1)
Faecaloma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric fistula (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric haemorrhage (Gastrointestinal disorders) | 3 (3) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 4 (4) | 4 (5)
Gastrointestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 3 (3)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 2 (2)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 5 (5) | 7 (7)
Oesophageal fistula (Gastrointestinal disorders) | 2 (2) | 0 (0)
Oesophageal obstruction (Gastrointestinal disorders) | 5 (5) | 3 (3)
Oesophageal stenosis (Gastrointestinal disorders) | 1 (1) | 4 (4)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pneumatosis intestinalis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 4 (4) | 5 (5)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 4 (4) | 6 (6)
Vomiting (Gastrointestinal disorders) | 9 (11) | 6 (7)
Asthenia (General disorders) | 2 (2) | 1 (1)
Chest discomfort (General disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1)
Death (General disorders) | 2 (2) | 7 (7)
Fatigue (General disorders) | 3 (3) | 6 (6)
General physical health deterioration (General disorders) | 1 (1) | 1 (1)
Malaise (General disorders) | 1 (1) | 0 (0)
Mucosal inflammation (General disorders) | 1 (1) | 4 (4)
Multiple organ dysfunction syndrome (General disorders) | 1 (1) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (2)
Pneumatosis (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 5 (8) | 1 (1)
Strangulated hernia (General disorders) | 1 (2) | 0 (0)
Sudden cardiac death (General disorders) | 1 (1) | 0 (0)
Systemic inflammatory response syndrome (General disorders) | 1 (1) | 0 (0)
Vascular device occlusion (General disorders) | 0 (0) | 1 (1)
Autoimmune hepatitis (Hepatobiliary disorders) | 2 (2) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 1 (1) | 0 (0)
Biliary obstruction (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis chronic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Granulomatous liver disease (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 2 (2) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Liver disorder (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Abdominal infection (Infections and infestations) | 1 (1) | 0 (0)
Abdominal wall infection (Infections and infestations) | 0 (0) | 1 (1)
Abscess (Infections and infestations) | 1 (1) | 0 (0)
Acute sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Anal abscess (Infections and infestations) | 1 (1) | 1 (2)
Bacteraemia (Infections and infestations) | 2 (2) | 2 (2)
Bronchitis (Infections and infestations) | 2 (2) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 1 (2) | 1 (1)
Cytomegalovirus infection (Infections and infestations) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 3 (4) | 0 (0)
Device related sepsis (Infections and infestations) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1)
Extradural abscess (Infections and infestations) | 0 (0) | 1 (1)
Gastrointestinal bacterial infection (Infections and infestations) | 0 (0) | 1 (1)
Giardiasis (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 1 (1)
Intervertebral discitis (Infections and infestations) | 0 (0) | 1 (1)
Large intestine infection (Infections and infestations) | 0 (0) | 1 (1)
Oral candidiasis (Infections and infestations) | 0 (0) | 1 (1)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 38 (40) | 32 (36)
Pneumonia aspiration (Infections and infestations) | 11 (11) | 7 (8)
Pneumonia influenzal (Infections and infestations) | 1 (1) | 0 (0)
Psoas abscess (Infections and infestations) | 0 (0) | 1 (1)
Pulmonary sepsis (Infections and infestations) | 3 (3) | 0 (0)
Pulmonary tuberculosis (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Salmonellosis (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (2) | 5 (5)
Septic shock (Infections and infestations) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 1 (1)
Stoma site infection (Infections and infestations) | 1 (1) | 1 (1)
Systemic candida (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Vascular device infection (Infections and infestations) | 1 (1) | 0 (0)
Viral myositis (Infections and infestations) | 1 (1) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Anastomotic fistula (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Gastrointestinal anastomotic stenosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Gastrostomy tube site complication (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Product administration error (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tracheal haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tracheal obstruction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 3 (3) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 2 (2)
Blood creatinine increased (Investigations) | 3 (3) | 2 (2)
Neutrophil count decreased (Investigations) | 4 (4) | 6 (7)
Platelet count decreased (Investigations) | 5 (5) | 10 (13)
White blood cell count decreased (Investigations) | 2 (2) | 4 (4)
Cachexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 6 (6) | 6 (6)
Dehydration (Metabolism and nutrition disorders) | 6 (6) | 8 (9)
Hyperammonaemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (3)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypochloraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 7 (7) | 6 (6)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 7 (8) | 6 (6)
Hypophagia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypovolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Malnutrition (Metabolism and nutrition disorders) | 2 (4) | 3 (3)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gastrointestinal submucosal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Neoplasm swelling (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 1 (1) | 3 (3)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 2 (2) | 3 (3)
Cognitive disorder (Nervous system disorders) | 1 (1) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 1 (1) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 1 (1)
Loss of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 1 (1)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0)
Vocal cord paralysis (Nervous system disorders) | 0 (0) | 1 (1)
Device dislocation (Product Issues) | 1 (1) | 0 (0)
Device failure (Product Issues) | 1 (1) | 0 (0)
Device occlusion (Product Issues) | 1 (1) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1) | 3 (3)
Personality change (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 11 (12) | 6 (6)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 0 (0)
Prerenal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 3 (4)
Renal impairment (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal tubular necrosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 (0) | 1 (1)
Ureteric obstruction (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Oesophagobronchial fistula (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 12 (13) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 7 (7)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Tracheal stenosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cold sweat (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hospitalisation (Surgical and medical procedures) | 1 (1) | 0 (0)
Aortic thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 2 (2) | 3 (3)
Dry gangrene (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 2 (2) | 0 (0)
Jugular vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 0 (0) | 1 (1)
Subclavian vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Vena cava thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Venous thrombosis (Vascular disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab + SOC (N=370) | Placebo + SOC (N=370)
Anaemia (Blood and lymphatic system disorders) | 185 (288) | 199 (295)
Leukopenia (Blood and lymphatic system disorders) | 25 (56) | 29 (72)
Neutropenia (Blood and lymphatic system disorders) | 95 (190) | 90 (179)
Thrombocytopenia (Blood and lymphatic system disorders) | 28 (54) | 37 (57)
Tinnitus (Ear and labyrinth disorders) | 36 (38) | 27 (30)
Hyperthyroidism (Endocrine disorders) | 19 (19) | 3 (4)
Hypothyroidism (Endocrine disorders) | 40 (46) | 24 (27)
Abdominal pain (Gastrointestinal disorders) | 28 (33) | 18 (21)
Abdominal pain upper (Gastrointestinal disorders) | 20 (21) | 27 (41)
Constipation (Gastrointestinal disorders) | 147 (238) | 149 (210)
Diarrhoea (Gastrointestinal disorders) | 129 (226) | 120 (190)
Dysphagia (Gastrointestinal disorders) | 46 (56) | 53 (66)
Nausea (Gastrointestinal disorders) | 245 (523) | 231 (507)
Stomatitis (Gastrointestinal disorders) | 97 (160) | 93 (146)
Vomiting (Gastrointestinal disorders) | 121 (226) | 114 (200)
Asthenia (General disorders) | 58 (103) | 44 (71)
Chest pain (General disorders) | 28 (39) | 20 (21)
Fatigue (General disorders) | 147 (231) | 122 (182)
Malaise (General disorders) | 45 (75) | 42 (63)
Mucosal inflammation (General disorders) | 59 (114) | 65 (116)
Oedema (General disorders) | 22 (59) | 20 (50)
Oedema peripheral (General disorders) | 16 (20) | 29 (34)
Pyrexia (General disorders) | 53 (72) | 44 (60)
Pneumonia (Infections and infestations) | 20 (21) | 22 (23)
Upper respiratory tract infection (Infections and infestations) | 19 (19) | 18 (19)
Urinary tract infection (Infections and infestations) | 12 (15) | 23 (26)
Alanine aminotransferase increased (Investigations) | 24 (43) | 26 (32)
Aspartate aminotransferase increased (Investigations) | 25 (43) | 27 (33)
Blood creatinine increased (Investigations) | 78 (130) | 77 (115)
Lymphocyte count decreased (Investigations) | 24 (52) | 21 (47)
Neutrophil count decreased (Investigations) | 138 (279) | 107 (235)
Platelet count decreased (Investigations) | 59 (100) | 57 (96)
Weight decreased (Investigations) | 87 (97) | 89 (110)
White blood cell count decreased (Investigations) | 96 (215) | 67 (154)
Decreased appetite (Metabolism and nutrition disorders) | 162 (283) | 138 (239)
Dehydration (Metabolism and nutrition disorders) | 27 (32) | 25 (25)
Hyperglycaemia (Metabolism and nutrition disorders) | 18 (25) | 19 (29)
Hyperkalaemia (Metabolism and nutrition disorders) | 26 (47) | 29 (42)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 34 (43) | 49 (69)
Hypocalcaemia (Metabolism and nutrition disorders) | 27 (34) | 19 (25)
Hypokalaemia (Metabolism and nutrition disorders) | 64 (107) | 68 (109)
Hypomagnesaemia (Metabolism and nutrition disorders) | 34 (43) | 23 (29)
Hyponatraemia (Metabolism and nutrition disorders) | 63 (95) | 72 (108)
Hypophosphataemia (Metabolism and nutrition disorders) | 20 (27) | 22 (25)
Arthralgia (Musculoskeletal and connective tissue disorders) | 30 (38) | 24 (26)
Back pain (Musculoskeletal and connective tissue disorders) | 27 (34) | 30 (35)
Dizziness (Nervous system disorders) | 36 (42) | 30 (38)
Dysgeusia (Nervous system disorders) | 39 (46) | 32 (35)
Headache (Nervous system disorders) | 30 (56) | 25 (30)
Neuropathy peripheral (Nervous system disorders) | 37 (41) | 37 (43)
Peripheral sensory neuropathy (Nervous system disorders) | 36 (36) | 30 (32)
Insomnia (Psychiatric disorders) | 49 (59) | 44 (56)
Cough (Respiratory, thoracic and mediastinal disorders) | 59 (71) | 56 (64)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 34 (39) | 29 (29)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 56 (112) | 53 (102)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 19 (21) | 12 (12)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 22 (27) | 24 (24)
Alopecia (Skin and subcutaneous tissue disorders) | 55 (55) | 39 (40)
Dry skin (Skin and subcutaneous tissue disorders) | 20 (21) | 10 (10)
Pruritus (Skin and subcutaneous tissue disorders) | 31 (33) | 12 (13)
Rash (Skin and subcutaneous tissue disorders) | 44 (56) | 26 (33)
Hypertension (Vascular disorders) | 23 (24) | 29 (35)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results. Sponsor review can be expedited to meet publication timelines.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-10-17): https://cdn.clinicaltrials.gov/large-docs/19/NCT03189719/Prot_SAP_002.pdf